CLINICAL TRIAL: NCT04407429
Title: Vienna Versus SARS-CoV-2 Virus: A Prospective Large-scale Antibody Study of SARS-CoV-2 in Patients and Health Care Workers
Brief Title: Vienna Versus SARS-CoV-2 Virus Study
Acronym: VIVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christian Hengstenberg, Univ.-Prof., Medical University of Vienna
Other Study IDs: EK 1387/2020
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: SARS-CoV-2; COVID-19
Keywords: COVID-19; SARS-CoV-2; Immunity; Antibodies; Virus; Respiratory Virus; Immunoglobulins
MeSH Terms: conditions — COVID-19; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health care workers: Physicians, Nursing staff, Midwives, Medical-technical assistants (including medical, therapeutic and diagnostic healthcare staff, and medical and nursing assistants), administrative personnel with patient contact
  Interventions: Diagnostic Test: Laboratory Analyses
- Patients: Patients admitted for non-COVID related symptoms to the Vienna General Hospital with available residual serum samples.
  Interventions: Diagnostic Test: Laboratory Analyses

INTERVENTIONS:
Diagnostic Test: Laboratory Analyses — Storage of serum for SARS-CoV-2-antibodies and biomarkers

SUMMARY:
This study examines the seroprevalence against SARS-CoV-2 in health care workers and patients at the Vienna General Hospital.

DETAILED DESCRIPTION:
This study consists of 2 parts: a longitudinal study enrolling 3,000 health care professionals at the Vienna General Hospital testing their antibody status 6 times over a period of 12 months (Cohort A), and a serial cross-sectional study of 3,000 patients (i.e., a total of 9,000 patients) admitted to the Vienna General Hospital for non-COVID-19-related symptoms at 3 different time points during this pandemic (Cohort B).

ELIGIBILITY:
Cohort A:

Inclusion criteria:

* Physicians
* Nursing staff
* Midwives
* Medical-technical assistants (including medical, therapeutic and diagnostic healthcare staff, and medical and nursing assistants)
* Administrative personnel with patient contact

Exclusion Criteria:

* Not employed at the Medical University of Vienna or the Vienna General Hospital
* No signed informed consent

Cohort B:

Inclusion Criteria:

● Patients with available residual serum samples

Exclusion Criteria:

● Serum samples from COVID-19 triage units at the Vienna General Hospital

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cohort A: Health care workers
  Cohort B: Patients admitted for non-COVID related symptoms
Sampling Method: Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-06-27 (Estimated); Study Completion 2021-06-27 (Estimated)

PRIMARY OUTCOMES:
Prevalence of antibody status in healthcare workers and in patients admitted for non-COVID-19 related symptoms over time | 1 year

SECONDARY OUTCOMES:
Incidence rate of sero-conversion | 1 year
Identification of risk markers/factors for SARS-CoV-2 infection | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hengstenberg, Univ.-Prof., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Riesenhuber M, Nitsche C, Binder CJ, Schernhammer ES, Stamm T, Jakse F, Anwari E, Hamidi F, Haslacher H, Perkmann T, Hengstenberg C, Zelniker TA. Comparison of the prevalence of SARS-CoV-2 nucleoprotein antibodies in healthcare workers and an unselected adult and paediatric all-comer patient population: insights from a longitudinal study of healthcare workers and concurrent serial cross-sectional studies of patients at an academic medical centre in Austria. BMJ Open. 2023 Jan 18;13(1):e063760. doi: 10.1136/bmjopen-2022-063760. PMID 36657754